CLINICAL TRIAL: NCT03382990
Title: The Impacts of Different Stent Types in Acute Myocardial Infarction on the Risk of Atrial Fibrillation
Brief Title: Stent Placement and the Risk of New-onset AF in Patients With AMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Stent-AF Trial
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation New Onset; Acute Myocardial Infarction
Keywords: Atrial fibrillation; Acute myocardial infarction; Drug-eluting stent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- STEMI: Patients with STEMI treated with PCI and stent placement (DES or BMS)
  Interventions: Device: DES or BMS
- NSTEMI: Patients with NSTEMI treated with PCI and stent placement (DES or BMS)
  Interventions: Device: DES or BMS

INTERVENTIONS:
Device: DES or BMS — DES or BMS placement during the procedure of PCI in patients with AMI is depend on the operator's decision.

SUMMARY:
The benefit of a drug-eluting stent (DES) in patients with acute myocardial infarction (AMI) is controversial. This study will aim to observe the effect of a DES on the risk of new-onset AF in patients with AMI.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is the leading cause of mortality in the world. Early invasive strategy with percutaneous coronary intervention (PCI) has been demonstrated to be the most effective strategy to treat AMI. Although drug-eluting stent (DES) has not shown benefits to reduce mortality rate among AMI patients compared with bare-metal stent (BMS), the use of DES in real-world is increasing because of reduced restenosis rates. AMI patients are at higher risk to develop atrial fibrillation (AF) than general population. However, whether early PCI with DES implantation is related to a reduced risk of AF still remains unclear. The purpose of this study is to investigate the association of DES implantation and the risk of AF among patients with AMI treated by early PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled by primary diagnostic coding as acute myocardial infarction and treatment coding as receiving PCI between 2007 and 2013 in Taiwan National Health Insurance Research Database (NHIRD)

Exclusion Criteria:

1. Less than 20-years-old; Unknown sex and age
2. Not residents in Taiwan
3. Died during AMI admission
4. Previous history of AF
5. Receiving coronary artery bypass grafting (CABG), ventricular assist device (VAD), extracorporeal membrane oxygenation (ECMO), and heart transplantation during observational and/or database period
6. No stent implantation during PCI
7. Unknown stent types

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within the retrospective cohort, we include patients who had received a primary diagnosis of AMI based on the discharge claim between 2007 and 2013. After the exclusion by the mentioned criteria, patients with AMI treated with PCI and stent placement are intended to be analyzed in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
new-onset atrial fibrillation | one year
  new record or diagnostic claims of atrial fibrillation after hospital discharge from acute myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Li-Nien Chien, PhD, Study Chair — Taipei Medical University

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.